CLINICAL TRIAL: NCT02689037
Title: Angioplasty and Stenting for Patients With Symptomatic Intracranial Atherosclerosis: Study Protocol of a Randomized Controlled Trial
Brief Title: Angioplasty and Stenting for Patients With Symptomatic Intracranial Atherosclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The 476th Hospital of People's Liberation Army (Other)
Responsible Party: Principal Investigator, Feng-Feng Shen, Doctor, The 476th Hospital of People's Liberation Army
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12MA100
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — Angioplasty; Stents; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stenting+medical treatment (Experimental): Patients in PTAS+MT group will receive Percutaneous transluminal angioplasty and stenting and medical treatment (aspirin 100mg daily and clopidogrel 75mg daily)
  Interventions: Procedure: Percutaneous transluminal angioplasty and stenting; Drug: Aspirin plus clopidogrel
- Aspirin plus clopidogrel (Active Comparator): Patients in aspirin plus clopidogrel group will receive aspirin 100mg daily and clopidogrel 75mg daily for 90 days.
  Interventions: Drug: Aspirin plus clopidogrel

INTERVENTIONS:
Procedure: Percutaneous transluminal angioplasty and stenting — Surgeons will plant stents after vascular angioplasty in target ICAS vessels within 5 days after randomization.
  Other Names: PTAS
  Arms: stenting+medical treatment
Drug: Aspirin plus clopidogrel — aspirin 100mg daily and clopidogrel 75mg daily for 90 days
  Other Names: Aspirin+clopidogrel

SUMMARY:
Background: Effectiveness of Percutaneous transluminal angioplasty and stenting (PTAS) on prevention of events of stroke and death in patients with symptomatic intracranial atherosclerosis (ICAS) is controversial.

Aim: to determine whether PTAS plus medical treatment (MT) are superior to MT alone in preventing events of stroke and death in patients with symptomatic ICAS.

Methods: The investigators will carry out a randomized controlled trial in 3 hospitals in China. A total of 198 patients with ICAS will be randomized into 2 groups: PTAS+MT and MT group. All patients will receive aspirin (100 mg daily) and clopidogrel (75 mg daily) immediately after randomization, and patients in PTAS+MT group will receive surgery within 5 days after randomization. The patients will be followed up for 1 year after randomization and assessed for events of stroke and death at 30 days and 1 year after randomization, the incidence of recurrent ischaemic stroke in the stenting-involved vascular territory at 30 days and 1 year after randomization, incidence of in-stent restenosis at 1 year after randomization,etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years.
* Complaints of a Symptomatic ICAS: a history of recurrent transient ischemic attacks or an ischemic stroke within 1 year owing to a 70%-99% stenosis in an internal carotid artery, middle cerebral artery, vertebral artery, or basilar artery.
* A length ≤ 15mm of a stenosis in the target vessel and a vessel size >2.5mm.
* Hypoperfusion in the territory of the target vessels, which is determined by CT or MRI in 14 days before stenting.
* CT or MRI scans show no massive cerebral infarction (beyond half of the territory of middle cerebral artery (MCA)), intracranial hemorrhage, epidural or sub-dural hemorrhage, and intracranial brain tumor.
* Patients who understand the purpose of the study and have provided informed consent.

Exclusion Criteria:

* Not able to receive general anesthesia.
* Not able to receive angiographic assessment.
* A stenosis >50% in an extracranial carotid or vertebral artery on the ipsilateral side.
* Infarctions due to the perforators occlusion (determined by MRI scan), which is defined as basal ganglia or brainstem/thalamus infarction related with middle cerebral artery or basilar artery stenosis.
* A high risk (leading to a stroke or death) to deliver the stent to the lesion.
* A previous stent or angioplasty in the target lesion.
* Progressive neurological signs within 24 hours before enrolment
* Any haemorrhagic infarct within 14 days before enrolment
* The presence of a cardiac source of embolus
* Thrombolytic therapy within 24 hours before enrollment
* Presence of intraluminal thrombus proximal to or at the target lesion
* Myocardial infarction within previous 30 days
* Non-atherosclerotic lesions: arterial dissection, moya-moya disease; vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid pleocytosis; radiation-induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process, and suspected recanalized embolus.
* Known contraindications for aspirin and clopidogrel treatment.
* An modified Rankin scale≥3.
* With a childbearing potential or a positive pregnancy test in 1 week before enrolment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with events of stroke or death | at 30 days after randomization

SECONDARY OUTCOMES:
the incidence of recurrent ischaemic stroke in the stenting-involved vascular territory | 30 days and 1 year after randomization
neurological functional outcome by the Chinese version of National Institutes of Health Stroke Scale (C-NIHSS) | 30 days and 1 year after randomization
Proportion of patients with adverse events | 30 days and 1 year after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hang Lin, MD, Principal Investigator — Fuzhou General Hospital of Nanjing Command, People's Liberation Army and Clinical Medical College of Fujian Medical University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui XP, Lin M, Mu JS, Ye JX, He WQ, Fu ML, Li H, Fang JY, Shen FF, Lin H. Angioplasty and stenting for patients with symptomatic intracranial atherosclerosis: study protocol of a randomised controlled trial. BMJ Open. 2016 Nov 15;6(11):e012175. doi: 10.1136/bmjopen-2016-012175. PMID 27852711